CLINICAL TRIAL: NCT00488163
Title: Pilot Study of Atomoxetine To Enhance COgnition In Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Joseph Friedman, Principal Investigator, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00131-03-1284
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Schizophrenia
Keywords: schizophrenia; cognition; atomoxetine; norepinephrine; dopamine
MeSH Terms: conditions — Schizophrenia | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomoxetine (Active Comparator): Atomoxetine 40 mg compounded into capsules.
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator): Inactive matching compounding of placebo capsules
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — Dose escalation from 40 mg to 50 mg of Atomoxetine active treatment.
  Other Names: Strattera®

SUMMARY:
Relationships between altered prefrontal cortical dopamine, norepinephrine and some cognitive impairments of schizophrenia supports and approach for pharmacological remediation of cognitive symptoms through manipulations of prefrontal cortical dopamine and norepinephrine. Atomoxetine, a selective norepinephrine re-uptake inhibitor, produces a widespread increase in brain norepinephrine and a secondary and selective increase in prefrontal dopamine. Given this, we are evaluating atomoxetine's cognitive effects in a pilot placebo controlled trial in patients with schizophrenia. Moreover, an fMRI investigation was undertaken to assess the neural mechanisms underlying the cognitive effects of atomoxetine.

DETAILED DESCRIPTION:
Participants carrying a diagnosis of schizophrenia and receiving treatment with one of the following antipsychotic medications are eleigible for participation: risperidone, olanzapine, quetiapine, aripirazole. Following consent, participants will be observed for 4 weeks to ensure stability of their symptoms. Following this, there will be baseline assessments of symptom severity, cognitive ability, functional ability and an fMRI scan. Following this, participants will be randomly assigned to receive treatment with 40 mg of atomoxetine or placebo daily during a double-blind parallel designed four week treatment period, following which the dose of atomoxetine will be increased to 40 mg twice day (or matching placebo) for an additional 4 weeks. The cognitive assessment battery and MRI will be repeated following 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be males and females between the ages of 18 and 65
2. In good general medical health
3. For patient subjects, a DSM-IV diagnosis of schizophrenia, any subtype
4. Currently in remission or with stable, unchanging residual symptoms
5. Receiving treatment with olanzapine, aripiprazole, risperidone, or quetiapine as their antipsychotic medication at a stable dose for a minimum of eight weeks.
6. Able to complete neurocognitive tests
7. Able to give informed consent. All subjects will be required to have at least an 8th grade reading level and/or a full-scale IQ of at least 85 as assessed by the Wide Range Achievement Test (WRAT).

Exclusion Criteria:

1. Recent history (within previous year) of serious suicide, homicide, or physical violence, or current suicidal or homicidal thoughts
2. Any axis I DSM-IV diagnosis in addition to schizophrenia or schizoaffective disorder except substance abuse in remission
3. History of severe head trauma, neurological disorder, or medical illness which may contribute to the subjects' psychiatric symptoms or cognitive impairment
4. Medical illness which requires taking any medication that has CNS activity which is known to impair cognition.
5. Untreated or unstable hypertension.
6. Coronary artery disease.
7. Receiving concomitant anticholinergic drugs, antidepressants or mood stabilizers. If patient subjects are receiving benzodiazepines, they must be short or intermediate acting (e.g. alprazolam, lorazepam) and must be held 48 hours prior to cognitive testing
8. Unable to give informed consent
9. History of developmental disorder or less than an eighth

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2007-04 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Composite score on the Brief Assessment of Cognition in Schizophrenia | 8 weeks
  Cognitive performance as measured by the BACS

SECONDARY OUTCOMES:
Brain activation measured by functional magnetic resonance imaging | 8 weeks
  Differences between changes in brain oxygenation level dependent imaging measures between placebo and Atomoxetine

CONTACTS AND LOCATIONS:
Overall Officials: Joseph I Friedman, MD, Principal Investigator — Pilgrim Psychiatric Center
Locations (2):
- United States (2):
  - Pilgrim Psychiatric Center, Brentwood, New York
  - Mount Sinai Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bymaster FP, Katner JS, Nelson DL, Hemrick-Luecke SK, Threlkeld PG, Heiligenstein JH, Morin SM, Gehlert DR, Perry KW. Atomoxetine increases extracellular levels of norepinephrine and dopamine in prefrontal cortex of rat: a potential mechanism for efficacy in attention deficit/hyperactivity disorder. Neuropsychopharmacology. 2002 Nov;27(5):699-711. doi: 10.1016/S0893-133X(02)00346-9. PMID 12431845